CLINICAL TRIAL: NCT00357331
Title: A Randomized Placebo Controlled Double Blind Investigation of the Effects of Potassium Citrate on Bone Metabolism in Postmenopausal Osteopenia
Brief Title: The Effects of Potassium Citrate on Bone Metabolism
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0604008486
Record Dates: First submitted 2006-07-25; First posted 2006-07-27 (Estimated); Results first posted 2017-06-12 (Actual); Last update posted 2017-06-12 (Actual); Status verified 2017-05

CONDITIONS: Bone Diseases, Metabolic; Osteoporosis, Postmenopausal
Keywords: postmenopausal osteopenia; treatment; bone loss
MeSH Terms: conditions — Bone Diseases, Metabolic; Osteoporosis, Postmenopausal | interventions — Potassium Citrate

STUDY DESIGN:
Intervention Model Description: Double Blind Placebo Controlled Trial
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Potassium Citrate (Experimental): Potassium Citrate 20 meq twice daily
  Interventions: Drug: potassium citrate
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: potassium citrate

INTERVENTIONS:
Drug: potassium citrate — 20 meq by mouth in capsule form twice daily
  Other Names: uro cit

SUMMARY:
Skeletal buffering of chronic acid loads may contribute to a significant amount of bone loss over time. Evidence from a few small short-term studies suggests that basic compounds, namely potassium citrate and potassium bicarbonate may reduce bone loss and improve bone density.

The purpose of this study is to evaluate the effects of potassium citrate on bone metabolism. We hypothesize that administration of potassium citrate to postmenopausal women with osteopenia will reduce bone resorption and improve bone mineral density.

Postmenopausal women with osteopenia (T score between -1.0 and -2.5) and no history of fracture will be randomized to either daily potassium citrate or placebo for one year. Primary outcomes will be markers of bone turnover, which will be measured over 12 months. Secondary outcomes will be bone mineral density, compliance, and adverse events.

DETAILED DESCRIPTION:
Participants were recruited from a single academic center. Subjects underwent screening at the Clinical Translational Science Center (CTSC) at Weill Cornell Medical College (WCMC). Study visits occurred at the CTSC where investigators administered and monitored questionnaires, compliance, adverse events, and endpoint measurements. Subjects were assigned an anonymous study number at the beginning of the trial, which was used to track the participant's data throughout the study. The protocol was approved by the Institutional Review Board (IRB) and the procedures followed were in accordance with the ethical standards of the IRB and the CTSC. All patients provided informed consent.

Treatment Groups Participants were assigned to either the treatment or placebo group using a randomization schema generated by the statistician. The randomization method was blocked randomization with a blocking factor of 4. The blocked randomization was not stratified by any other factors. The study was conducted in a double blind manner. The study medication, K-citrate, or placebo, was dispensed through the New York Presbyterian Hospital (NYPH) pharmacy. Bottles in the pharmacy were sequentially numbered and the number was linked to the blocked randomization scheme. Only the statistician and the pharmacist knew the meaning of the numbered codes and only the statistician knew the blocking assignment. Blocked randomization with balanced randomization of each block and blocks of the same size was performed by the RANDOM procedure within the WinPepi Version 11.1.

Investigators who administered questionnaires and assessed compliance, adverse effects or endpoint information were blind to group assignment. Only study investigators were able to enroll participants in the study and assign them to treatment arms. Those assigned to the treatment group received the study drug (40 mEq daily K Citrate: two 10 mEq tablets twice daily); those assigned to the control group received inert tablets of the same quantity. All participants received daily supplementation with Citracal (630 mg calcium citrate and 400 IU vitamin D3 per two caplets). All supplements and medications were provided by Mission Pharmacal/Bayer Pharmaceuticals in Boerne, Texas. Subjects discontinued their prior supplements at the time of entry to the study and were advised to adhere to the standardized supplementation regimen outlined by the protocol.

Measurements and Outcomes Subjects were evaluated at baseline, 1, 3, 6, and 12 months. The following outcomes were measured: change in bone turnover markers including u-NTX, BSAP, OC and P1NP; changes in 24 hour urinary concentrations of citrate, sulfate, and calcium; and changes in BMD measured from baseline to 12 months. Adverse events and compliance were measured at each visit over the study duration. Adverse events pertained to medication side effects, including, but not limited to, gastrointestinal complaints, nausea, diarrhea, and stomach pain, as well as the development of hyperkalemia or metabolic acidosis. If any of the following occurred, potassium exceeded 5.2 mmol/L; bicarbonate level exceeded 32 mmol/L; creatinine increased by more than 30% or rose above 2.0 ng/dL; or GFR was < 60, study medications were stopped until the parameter normalized, at which point the medication was resumed at half dose: Compliance was assessed by remaining pill count; good compliance was defined at ≤ 20% of pills remaining, or ≤ 18 pills remaining for each 3-month dose allocation.

Baseline measurements included dietary assessment (block food frequency questionnaire) and blood pressure. Laboratory evaluation was performed at the General Core Laboratory at WCMC and included a basic metabolic panel, calcium, albumin and thyroid stimulating hormone (TSH). 25-OH and 1,25(OH)2 Vitamin D were measured by radioimmunoassay (Immunodiagnostic Systems, Scottsdale, Arizona). The interassay coefficient of variation (CV) was <8.2% and <13%, respectively. Intact parathyroid hormone (i-PTH) was measured by immunoradiometric assay (Scantibodies Laboratories, Santee, California; CV <6.4%). Markers of bone turnover included osteocalcin (OC: quantitative immunoradiometric assay, DiaSorin, Stillwater, Minnesota; CV <9.5%) , bone specific alkaline phosphatase (BSAP: solid phase monoclonal antibody immunoenzymetric assay, Immunodiagnostics Systems, Scottsdale, Arizona; CV<6.4%), procollagen type 1 amino-terminal propeptide (P1NP: quantitative radioimmunoassay, Orion Diagnostica, Espoo, Finland; CV<9.8%), urinary N-telopeptide (U-NTX: quantitative enzyme-linked immunosorbent assay kit, Wampole Laboratories INC Princeton, New Jersey; CV<5.0%). All specimens were collected as fasting morning samples. The urinary-NTX was a second morning void. The specimens were frozen and batch analyzed. 24 hour urinary collections for calcium, creatinine, sulfate, citrate and sodium were analyzed at Quest Diagnostics. BMD was performed at lumbar spine, total hip and femoral neck using dual-energy X-ray Absorptiometry (DXA) Hologic; Bedford, Massachusetts. The least significant change (LSC) for the DXA was 0.025 at the lumbar spine, 0.025 at the femoral neck and 0.015 at the radius. Two technologists, both certified by the International Society for Clinical Densitometry, performed all DXA testing on the participants.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women, more than 2 years post menopause
* Osteopenia, defined as a T score at the lumbar spine or total hip between -1.0 and -2.5
* No history of prior fragility fracture

Exclusion criteria:

* Renal insufficiency
* Use of potassium sparing diuretics
* Use of potassium supplements
* Hyperkalemia
* Secondary causes of osteoporosis or metabolic bone disease
* Delayed gastric emptying
* esophageal compression, intestinal obstruction or stricture
* use of anticholinergic medication
* active urinary tract infection.

Ages: 45 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2006-08 (Actual); Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Naina Sinha Gregory, M.D., Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gregory NS, Kumar R, Stein EM, Alexander E, Christos P, Bockman RS, Rodman JS. POTASSIUM CITRATE DECREASES BONE RESORPTION IN POSTMENOPAUSAL WOMEN WITH OSTEOPENIA: A RANDOMIZED, DOUBLE-BLIND CLINICAL TRIAL. Endocr Pract. 2015 Dec;21(12):1380-6. doi: 10.4158/EP15738.OR. Epub 2015 Sep 24. PMID 26401577

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo
  Placebo 20 meq by mouth in capsule form twice daily
Period: Overall Study
Arm/Group | Potassium Citrate | Placebo
Started | 42 | 41
Completed | 42 | 41
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Potassium Citrate | Total
Number analyzed (Participants) | 41 | 42 | 83
Age, Categorical [Count of Participants; unit: Participants]
  Age: <=18 years | 0 | 0 | 0
  Age: Between 18 and 65 years | 3 | 5 | 8
  Age: >=65 years | 38 | 37 | 75
Age, Continuous [Median (Standard Deviation); unit: years] | 66.1 (7.1) | 65.1 (5.9) | 65.8 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 42 | 83
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants] — New York City & Surrounding Environs
  participants
    United States | 41 | 42 | 83
BMI [Median (Standard Deviation); unit: kg/m2] | 23 (2.5) | 24 (3.3) | 23 (3.0)
PTH [Median (Standard Deviation); unit: pg/mL] | 58.8 (25) | 56.9 (33.4) | 57.2 (28)
25-OH Vitamin D [Median (Standard Deviation); unit: ng/mL] | 35.3 (12.7) | 31.3 (13.3) | 33.3 (13)

OUTCOME MEASURES:

1. Primary Outcome: Urinary-N-telopeptide
Description: One measure of bone turnover was urinary-NTX as a second void morning urine.
Time Frame: Baseline,1,3,6,12 months
Population: The numbers analyzed reflect the number of participants evaluable at each time point.
Measure: Mean (Standard Deviation); unit: nml BCE/nmol creatinine
Arm/Group | Placebo | Potassium Citrate
Number analyzed (Participants) | 39 | 37
nml BCE/nmol creatinine
  Baseline | 47.2 (19.6) | 51.6 (25.8)
  Month 1: number analyzed (Participants) | 32 | 35
  Month 1 | 44.5 (22.5) | 47 (21)
  Month 3: number analyzed (Participants) | 27 | 34
  Month 3 | 50.8 (21.2) | 40.5 (24.5)
  Month 6: number analyzed (Participants) | 27 | 29
  Month 6 | 40.4 (11.6) | 41.6 (18.4)
  Month 12: number analyzed (Participants) | 26 | 29
  Month 12 | 42.1 (13.9) | 41.6 (18.4)

2. Secondary Outcome: Number of Participants With Stable Bone Mineral Density (BMD) Over 12 Months at All Sites.
Description: BMD was performed at lumbar spine, total hip and femoral neck using dual-energy X-ray Absorptiometry (DXA) Hologic; Bedford, Massachusetts.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Potassium Citrate
Number analyzed (Participants) | 41 | 42
Participants | 41 | 42

3. Primary Outcome: P1NP (Amino-terminal Propeptide of Type I Procollagen)
Description: One measure of bone turnover was P1NP as a morning lab draw.
Time Frame: Baseline,1,3,6,12 months
Population: The numbers analyzed reflect the number of participants evaluable at each time point.
Measure: Mean (Standard Deviation); unit: micrograms/L
Arm/Group | Placebo | Potassium Citrate
Number analyzed (Participants) | 41 | 42
micrograms/L
  Baseline | 50.6 (20.1) | 55.5 (23.5)
  Month 1: number analyzed (Participants) | 35 | 36
  Month 1 | 48.9 (19.2) | 48.1 (16.9)
  Month 3: number analyzed (Participants) | 34 | 36
  Month 3 | 48.7 (18.3) | 43.5 (15.5)
  Month 6: number analyzed (Participants) | 31 | 33
  Month 6 | 46.0 (15.0) | 43.2 (12.8)
  Month 12: number analyzed (Participants) | 29 | 31
  Month 12 | 45.5 (16.5) | 42.4 (13.6)

ADVERSE EVENTS:
Arm/Group | Potassium Citrate | Placebo
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/41
Other Adverse Events (participants affected / at risk) | 10/42 | 11/41
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Potassium Citrate (N=42) | Placebo (N=41)
Traumatic Ankle Fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 2 | 6
Gastrointestinal Symptoms (Gastrointestinal disorders) | 8 | 4

LIMITATIONS AND CAVEATS:
Possible dual effect of calcium citrate, which mitigated the net effect of the alkalinizing treatment. The dose of K-citrate may not be sufficient to produce a change in BMD. Duration of treatment may have been too short to see changes in BMD.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No